CLINICAL TRIAL: NCT05407090
Title: The Effect of Probiotic Supplementation on Systemic Inflammation and Metabolic Endotoxemia in Morbidly Obese Patients Undergoing Bariatric Surgery
Brief Title: The Effect of Probiotics on Systemic Inflammation and Metabolic Endotoxemia in Patients Undergoing Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NKBBN/447/2021/MP
Record Dates: First submitted 2022-05-25; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Bariatric Surgery Candidate; Dysbiosis
Keywords: microbiota; bariatric surgery; obesity; inflammation; endotoxemia; intestinal permeability
MeSH Terms: conditions — Dysbiosis; Obesity; Inflammation; Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Patients will take 4 capsules of a multi-strain probiotic preparation daily. Product characteristics: 1 capsule of the preparation contains ≥2.5 x 10^9 CFU / g of live bacteria (Bifidobacterium lactis W52, Lactobacillus brevis W63, Lactobacillus casei W56, Lactococcus lactis W19, Lactococcus lactis W58, Lactobacillus acidophilus W37, Bifidobacterium bifidillum W23)
  Interventions: Dietary Supplement: probiotic supplementation
- Placebo (Placebo Comparator): Patients will take 4 capsules of a placebo preparation daily.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotic supplementation — Participants enrolled in the probiotic group will receive probiotics for 12 weeks before surgery.
  Arms: Probiotic
Dietary Supplement: placebo — Participants enrolled in the placebo group will receive a placebo instead of probiotics.
  Arms: Placebo

SUMMARY:
This study explores the effects of probiotic administration on the outcomes of surgical treatment, and also on the state of the intestinal microbiota and the intestinal barrier. The study protocol is designed as a randomized double-blind placebo-controlled clinical trial. Patients qualified for bariatric surgery will be randomized to receive probiotics or a placebo for 12 weeks. Researchers are going to evaluate changes in intestinal microbiota, epithelial permeability, weight loss, postoperative complications, and serum parameters reflecting inflammation, metabolic profile, and metabolic endotoxemia.

DETAILED DESCRIPTION:
The study is designed as a randomized double-blind placebo-controlled clinical trial with a 12-week probiotics intervention period. Eighty patients qualified for one of 3 types of bariatric surgery Roux-en-Y Gastric Bypass (RYGB), One-Anastomosis Gastric Bypass (OAGB), Laparoscopic Sleeve Gastrectomy (LSG) will be randomized to receive probiotics or a placebo. The time frame for the study is 6 months before and 6 months after surgery.

During this time, it is planned to collect stool samples at 5-time points: before the start of the study, before the introduction of probiotic therapy, 2 weeks before the operation, and 3 and 6 months after the operation. Collected fecal samples will be subjected to quantitative and qualitative content of the intestinal microbiota using the new generation sequencing method, as well as intestinal permeability parameters such as I-FABP (Intestinal fatty acid-binding protein), bacterial short-chain fatty acids (SCFA), and lipopolysaccharide (LPS).

Simultaneously with the collection of stool samples, an assessment of the patient's nutrition will be performed using the food frequency questionnaire (FFQ) and three-day dietary recall.

The blood samples will be collected at 4-time points: before the start of the study, before the operation, and 3 and 6 months after the operation. The following parameters will be marked in the collected blood samples: glucose, insulin, HbA1c, liver tests: ALT (Alanine transaminase), AST (Aspartate transaminase), GGTP (Gamma-glutamyl Transferase), alkaline phosphatase (ALP), bilirubin; lipid profile, CRP (C-reactive protein), total protein, albumin, inflammatory markers: IL-6, IL-10, Tumor necrosis factor-α (TNF-α), IL-8, IL-R2.

During the examination, tissue samples will be taken at 2-time points. The first is during routine gastroscopy before surgery. Gastroscopy will be performed before the inclusion of the probiotic. Duodenal and stomach biopsy will be performed during gastroscopy. The second time tissue samples will be collected intraoperatively. Gastric specimens will be collected from patients undergoing LSG. Patients qualified for RYGB and OAGB surgery will undergo gastric and jejunum biopsy. The parameters of the intestinal barrier status will be assessed in the collected tissues: Plasmalemma Vesicle-Associated Protein-1 (PLVAP-1), and Regenerating Islet Derived Protein 3 Alpha (Reg3α).

ELIGIBILITY:
Inclusion Criteria:

* qualification for LSG, RYGB, OAGB bariatric surgery
* age over 18
* written consent to participate in the study

Exclusion Criteria:

* allergy/intolerance to any of the ingredients of the preparations,
* inflammatory bowel diseases,
* current antibiotic therapy,
* immunosuppression,
* biological treatment,
* long-term antibiotic therapy,
* taking probiotics in the 1 month prior to study enrollment,
* neurodegenerative diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of changes in weight loss of the body | 3 and 6 months after surgery
  Weight loss will be measured and expressed in kilograms
Evaluation of changes in inflammation status | before the intervention, 3 and 6 months after surgery
  The inflammation will be assessed by measuring CRP concentration in the serum

SECONDARY OUTCOMES:
Evaluation of changes in the state of the intestinal microbiota - the content of intestinal microbiota | before the intervention, 2 weeks before surgery, 3 and 6 months after surgery
  The state of the intestinal microbiota will be measured by quantitative and qualitative content of the intestinal microbiota using the new generation sequencing method (16s rRNA)
Evaluation of changes in the state of the intestinal microbiota - the content of bacterial metabolites short-chain fatty acids (SCFA) | before intervention, 2 weeks before surgery, 3 and 6 months after surgery
  The state of the intestinal microbiota will be measured by the quantitative and qualitative content of bacterial metabolites - short-chain fatty acids (SCFA)
Evaluation of changes in the permeability of the intestinal barrier | before the intervention, 2 weeks before surgery, 3 and 6 months after surgery
  The permeability of the intestinal barrier will be measured by the presence of increased intestinal permeability parameter - I-FABP in stool
Evaluation of changes in the state of the intestinal barrier | before the intervention, in time of surgery
  The permeability of the intestinal barrier will be measured by the concentration of PLVAP-1 and Reg3-alfa in collected tissues
Evaluation of changes in endotoxemia | before the intervention, 3 and 6 months after surgery
  Endotoxemia will be assessed by measuring lipopolysaccharide in serum.
Evaluation of changes in inflammation profile in serum | before the intervention, 3 and 6 months after surgery
  The inflammation profile will be assessed by a concentration of cytokines (IL-6, TNF-alfa, IL-10, IL-8, IL-2R) in the serum.
Evaluation of changes in intestine inflammation | before the intervention, 3 and 6 months after surgery
  The intestine inflammation will be measured by the level of calprotectin in the stool
Evaluation of changes in nutrition - frequency | before the intervention and 6 months after surgery
  The assessment of the nutrition will be performed using the food frequency questionnaire (FFQ)
Evaluation of changes in nutrition - quality and quantity | two weeks before surgery and 3 months after surgery
  The assessment of the nutrition will be performed using a 3-day food record
Postoperative complications | During six months after surgery
  Postoperative complications will be assessed by the Clavien-Dindo classification of surgical complications (on a scale of 1 to 5, the higher the result, the more intensive treatment is required for the described complication)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Potrykus, Principal Investigator — Department of General, Endocrine and Transplant Surgery, Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk, Gdansk, Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potrykus M, Stanislawowski M, Czaja-Stolc S, Potrykus A, Stankiewicz M, Owczarzak A, Guzek M, Szymanski M, Loniewski I, Adrych K, Malgorzewicz S, Kaska L, Slebioda T, Proczko-Stepaniak M. 12-week preoperative probiotic supplementation versus placebo: effects on inflammation, endotoxemia, adipokines, and gastrointestinal peptides in patients six months after bariatric surgery - a double-blind, randomized, placebo-controlled clinical trial. Nutr J. 2025 Oct 9;24(1):156. doi: 10.1186/s12937-025-01217-2. PMID 41068905